CLINICAL TRIAL: NCT05170217
Title: Reducing the Harmful Effects of Cannabis Use: Finding the Optimal CBD:THC Ratio
Acronym: eCBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HR-16/17-4163
Record Dates: First submitted 2021-11-17; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-11

CONDITIONS: Cannabis Use
MeSH Terms: interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CBD:THC 0:1 (Experimental): Inhalation of cannabis containing only THC
  Interventions: Drug: THC
- CBD:THC 1:1 (Experimental): Inhalation of cannabis containing THC and CBD
  Interventions: Drug: THC; Drug: Cannabidiol
- CBD:THC 2:1 (Experimental): Inhalation of cannabis containing THC and CBD
  Interventions: Drug: THC; Drug: Cannabidiol
- CBD:THC 3:1 (Experimental): Inhalation of cannabis containing THC and CBD
  Interventions: Drug: THC; Drug: Cannabidiol

INTERVENTIONS:
Drug: THC — Inhaled cannabis containing 10mg THC
Drug: Cannabidiol — Inhaled cannabis containing 10mg CBD
  Arms: CBD:THC 1:1
Drug: Cannabidiol — Inhaled cannabis containing 20mg CBD
  Arms: CBD:THC 2:1
Drug: Cannabidiol — Inhaled cannabis containing 30mg CBD
  Arms: CBD:THC 3:1

SUMMARY:
This study will recruit healthy volunteers who use cannabis infrequently. Each participant will attend the laboratory on five occasions: an initial visit to check that they are safe to join the study and four days of testing.

Participants will be administered, in a randomized order, vaporized cannabis containing one of four different ratios of CBD:THC (0:1, 1:1, 2:1, 3:1). The cannabis administration will follow a standardised inhalation procedure using a medical-grade vaporizer device.

Participants will complete a series of tasks measuring cognition, psychosis, anxiety and other subjective experiences.

The study will be carried out at the NIHR-Wellcome Trust Clinical Research Facility at King's College Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Female and male volunteers aged 21-50
* Have used cannabis at least once
* Willing to provide written informed consent
* Willing to provide blood samples
* Fluent English speaker

Exclusion Criteria:

* Past or present major mental illness
* Past or present major physical illness
* Past or present substance use disorder
* Past or present use of anti-psychotic or anti-depressant medications
* First degree relative with psychotic disorder
* Currently taking psychotropic medication
* Positive urine drug screen at screening or experimental visits
* Use of alcohol 24h prior to experimental visit or tobacco on the day of experiment
* Pregnancy (current or planned) or lactation in women
* Significant abnormality detected during physical examination at screening visit
* Cannabis use (defined as days in which cannabis is used recreationally) more than once per week on average over the last 12 months
* Any past use of synthetic cannabinoids
* Score of 5 and above on the Fagerstrom Nicotine dependence questionnaire
* BMI classified as obese or underweight
* Taken part in any drug study within the last 30 days or taking part in another study over the course of the trial
* Known drug sensitivity/allergy towards cannabis or Lorazepam

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-06-09 (Actual); Study Completion 2019-06-09 (Actual)

PRIMARY OUTCOMES:
Hopkins Verbal Learning Task | 40-45 minutes post cannabis inhalation
  Delayed verbal recall

SECONDARY OUTCOMES:
Hopkins Verbal Learning Task | 20-40 minutes post cannabis inhalation
  Immediate verbal recall
Forward and Reverse Digit span | 20-40 minutes post cannabis inhalation
  Working memory
Spatial N-back task | 20-40 minutes post cannabis inhalation
  Spatial working memory
Positive and Negative Syndrome Scale | Baseline; 3-4 hours post cannabis inhalation
  Positive subscale
State Social Paranoia Scale | 3-4 hours post cannabis inhalation
Community assessment of Psychic Experiences - state | 3-4 hours post cannabis inhalation
Psychotomimetic states inventory | 3-4 hours post cannabis inhalation
Visual analogue scales (0 to 100 millimetres) | Baseline; Pre-cannabis, 10 minutes post-cannabis, 50 minutes post-cannabis, 1 hour 10 minutes post-cannabis, discharge
  * Feel drug effect
  * Like drug effect
  * Want more drug
  * Mentally impaired
  * Dry Mouth
  * Enhanced colour perception
  * Enhanced sound perception
  * Want food
  * Want alcohol
  * Feel high
  * Feel anxious
  * Feel paranoid
  * Feel tired
  * Feel calm and relaxed
  * Feel stoned
  * The drug effects are pleasurable
Pleasurable responses - Visual analogue scale (-50 to 50 millimetres) | 1 hour post-cannabis
  Increased or decreased pleasure from chocolate and music during intoxication
Plasma THC concentration | Pre-cannabis, 0 minutes post-cannabis, 5 minutes post-cannabis, 15 minutes post-cannabis, 90 minutes post-cannabis
Plasma CBD concentration | Pre-cannabis, 0 minutes post-cannabis, 5 minutes post-cannabis, 15 minutes post-cannabis, 90 minutes post-cannabis
Plasma 11-OH-THC concentration | Pre-cannabis, 0 minutes post-cannabis, 5 minutes post-cannabis, 15 minutes post-cannabis, 90 minutes post-cannabis
Plasma 11-COOH-THC concentration | Pre-cannabis, 0 minutes post-cannabis, 5 minutes post-cannabis, 15 minutes post-cannabis, 90 minutes post-cannabis
Plasma 7-OH-CBD concentration | Pre-cannabis, 0 minutes post-cannabis, 5 minutes post-cannabis, 15 minutes post-cannabis, 90 minutes post-cannabis

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliver D, Englund A, Chesney E, Chester L, Wilson J, Sovi S, Wigroth S, Hodsoll J, Strang J, Murray RM, Freeman TP, Fusar-Poli P, McGuire P. Cannabidiol does not attenuate acute delta-9-tetrahydrocannabinol-induced attentional bias in healthy volunteers: A randomised, double-blind, cross-over study. Addiction. 2024 Feb;119(2):322-333. doi: 10.1111/add.16353. Epub 2023 Oct 11. PMID 37821096
- [Derived] Chester LA, Englund A, Chesney E, Oliver D, Wilson J, Sovi S, Dickens AM, Oresic M, Linderman T, Hodsoll J, Minichino A, Strang J, Murray RM, Freeman TP, McGuire P. Effects of Cannabidiol and Delta-9-Tetrahydrocannabinol on Plasma Endocannabinoid Levels in Healthy Volunteers: A Randomized Double-Blind Four-Arm Crossover Study. Cannabis Cannabinoid Res. 2024 Feb;9(1):188-198. doi: 10.1089/can.2022.0174. Epub 2022 Dec 9. PMID 36493386